CLINICAL TRIAL: NCT03127670
Title: Effect of Solanum Melongena Extract in the Treatment of Arsenical Skin Lesion
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bangabandhu Sheikh Mujib Medical University, Dhaka, Bangladesh (Other)
Responsible Party: Principal Investigator, Prof. Mir Misbahuddin, Professor, Bangabandhu Sheikh Mujib Medical University, Dhaka, Bangladesh
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BSMMU-012-CT
Record Dates: First submitted 2017-04-12; First posted 2017-04-25 (Actual); Last update posted 2018-07-13 (Actual); Status verified 2018-07

CONDITIONS: Arsenical Keratosis

STUDY DESIGN:
Intervention Model Description: Solanum melongena peel extract
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Solanum melongena peel extract 0.05% (Experimental): 25 Patients Solanum melongena peel extract 0.05% Twice daily applied topically for 12 weeks
  Interventions: Drug: Solanum melongena peel extract 0.05%

INTERVENTIONS:
Drug: Solanum melongena peel extract 0.05% — Administered topically twice daily for 12 weeks
  Other Names: Solanum melongena peel extract cream

SUMMARY:
Solanum melongena is a common vegetable contains phytochemicals which prevent, reduce or delay the oxidation of DNA and alter the cellular signal transduction pathways controlling cell proliferation and apoptosis of human cancer. The skin of Solanum melongena peel contains nasunin an anthocyanins and chlorogenic acid which have anti-inflammatory, antioxidant, antimutagenic and antiangiogenic properties. Extract of Solanum melongena is used in actinic keratosis and Squamous cell carcinoma of the skin. This study will determine any change in arsenical skin lesion after administrating Solanum melongena extract cream.

DETAILED DESCRIPTION:
Bangladesh is grappling with the world greatest ever environmental health disaster in history. About three decades, more than thirty millions people subsistence with this problem without any potential treatment. So, now arsenic crisis as a major issue and becomes a demand of era to find out the way to solve this problem. Chronic ingestion of arsenic contaminated water is a silent killer of the human because even it may cause death by carcinoma. Arsenic has an affinity to keratin-rich tissue like skin, hair, nail due to the presence of sulphydryl group, as a consequence, they manifest of clinical symptoms like hyperpigmentation or melanosis, diffuse dark brown spot of skin or characteristic rain drop appearance over the trunks, limbs; keratosis. Even due to prolong exposure to arsenic e.g. invasive skin lesion as Bown's disease and squamous cell carcinoma appear. Arsenic as neglected disease arsenic patients has no established treatment except preventive and supportive treatment of melanosis by drinking arsenic free water and salicylic acid as keratolytic substance. But the malignant condition of arsenic skin lesion treatment is not yet documented. Solanum melongena belongs to Leptostemonum Clade (the "spine" solanums) species-rice in solanaceae. It also called brinjal or eggplant. Solanum melongena is a common vegetable contains phytochemicals which prevent, reduce or delay the oxidation of DNA and alter the cellular signal transduction pathways controlling cell proliferation and apoptosis of human cancer. Polyphenols of Solanum melongena exhibit an anticancer effect both in vitro and in vivo experiments. Polyphenol reduces scavenge free radicals, induce apoptosis, inhibit cell proliferation and angiogenesis and exhibit phytoestrogen activity. On other hand, they suppress the NF-κB and the activating protein (AP-1), inhibit the mitogen-activated proteins (MAPKs), the protein kinase and growth factor receptor-mediated pathways which are involved in cell cycle arrest and possess anti-inflammatory properties. Solanum melongena has solasodine glycoalkaloids which are cytotoxic and bind with endogenous endocytic lectin of cancer cell membrane and induce apoptosis and cell death both in vivo and in vitro. The skin of Solanum melongena peel contains nasunin an anthocyanins and chlorogenic acid which have anti-inflammatory, antioxidant, antimutagenic and antiangiogenic properties. It has a cytotoxic effect on brine shrimp. Therefore, this study will be conducted to determine is there any change in the patient with arsenical skin lesions before and after application of topical Solanum melongena extract cream. Twenty-five patients with arsenical skin lesions will be recruited on the basis of inclusion and exclusion criteria after IRB approval. The patients will be applied Solanum melongena extract cream twice daily for 12 weeks without any interruption. Water and nails samples will be collected for confirming the diagnosis. Blood samples will be collected before and after treatment to evaluate the liver and renal function tests. So, this study will determine any change in arsenical skin lesion after administrating Solanum melongena extract cream.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18-60 years
* Sex: Both male and female
* Arsenicosis: Severe arsenical skin lesions with Bowen's disease or Squamous cell carcinoma
* Drinking arsenic contaminated water (> 50 µg/L) for more than 6 months
* Patient voluntarily agreed to participate
* Patient who understood the instruction of applying medicine and apply it as he or she will be instructed

Exclusion Criteria:

* Age: Less than 18 and above 60 years
* Expectant, Pregnant and lactating mother
* Major health problems Tuberculosis, Hepatic diseases, Renal diseases, Systamic lupus erythrometosis,
* Rheumatoid arthritis
* Patient with other skin diseases like ectopic dermatitis, psoriasis, eczema, drug allergy
* Food allergy of Solanum melongena
* Patient who received treatment within last three months
* Patient with Bowen disease and Squamous cell carcinoma due to other cause
* Patient did not voluntarily agree to participants

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2016-11-14 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2017-12-31 (Actual)

PRIMARY OUTCOMES:
Changes in palmer arsenical keratosis | Clinical outcome [Time Frame:[0 week (baseline),12 weeks (end)] [Safety Issue: No]] [Safety Issue: No]]
  Size of keratotic lesion will be decreased

SECONDARY OUTCOMES:
Changes in the liver function test | Change in lesion size [ Time Frame: [0 week (baseline), 12 weeks (end)] [Safety Issue: No]] [Safety Issue: No]]
  Abnormal liver function tests will be returned toward normal

CONTACTS AND LOCATIONS:
Overall Officials: Mir Misbahuddin, PhD, Study Director — Bangabandhu Sheikh Mujib Medical University, Dhaka, Bangladesh
Locations (1):
- Bhanga, Farīdpur, Bangladesh

IPD SHARING:
Plan to Share IPD: No